CLINICAL TRIAL: NCT05362578
Title: Wearable Transcutaneous Electrical Acustimulation for Gastroparesis
Brief Title: Transcutaneous Electrical Acustimulation (TEA) for Gastroparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Borko Nojkov, Clinical Lecturer - Specialty Gastroenterology, Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00204800; 5R44AT011380-02 (NIH)
Record Dates: First submitted 2022-03-31; First posted 2022-05-05 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Gastroparesis With Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Masking Description: Half of subjects will be randomized to the sham arm, and half will be randomized to the treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment group (Experimental): Subjects will be trained to use the devices at the treatment points and will undergo the treatment twice per day for 8 weeks. Following the first 8 weeks, at visit two, the devices will be collected by the study team.
  Interventions: Device: transcutaneous electrical accustimulation at treatment point.
- Sham group (Sham Comparator): Subjects will be trained to use the devices at sham points and will undergo sham stimulation for the first 8 weeks. At visit two, after unmasking, subjects will optionally be trained on the treatment points and may participate in treatment for 4 weeks.
  Interventions: Device: transcutaneous electrical accustimulation at sham point.

INTERVENTIONS:
Device: transcutaneous electrical accustimulation at treatment point. — The transcutaneous electrical accustimulator (TEA) device administers a mild electrical shock through the skin, similar to acupuncture at a location previously seen to provide benefit. The precise distinction between sham and experimental accustimulation is not described upon registration to reduce unblinding risk, to maintain scientific integrity.
  Arms: Treatment group
Device: transcutaneous electrical accustimulation at sham point. — The transcutaneous electrical accustimulator (TEA) device administers a mild electrical shock through the skin, similar to acupuncture at a location which has not been shown to provide benefit. The precise distinction between sham and experimental accustimulation is not described upon registration to reduce unblinding risk, to maintain scientific integrity.
  Arms: Sham group

SUMMARY:
The device being studied, the Transcutaneous Electrical Accustimulator (TEA), will deliver weak electrical current at two specific points, one at the leg and the other at the arm at settings known to improve symptoms involving the digestive system. The study team would like to test if the device will impact the gastrointestinal (GI) symptoms and gastric motility in study participants with gastroparesis.

DETAILED DESCRIPTION:
This study aims to assess if the device will impact the (GI) symptoms and gastric motility in study participants with gastroparesis. This will be done over a 12 week period during which each participant will undergo two visits. There will be two total visits that each follow the same schedule. During the first visit, subjects will undergo a 3-in-1 gastric functional test which is a non-invasive method to assess the gastric motility and visceral pain. This test will entail an EGG, ECG, and water satiety drink test for gastric accommodation. Following the 3-in-1 gastric functional test, subjects will be randomized and trained on how to use the study device. Half of the patients will be assigned to the sham group and half will be assigned to the treatment group. Each group will undergo 8 weeks of treatment or 8 weeks of sham stimulation and will receive weekly calls from the study team to check for adverse events and study compliance. Following the first 8 week period, subjects will return to the study site to undergo visit two. This will follow the same format as visit 1. At this time, subjects will become unblinded. Those who received sham stimulation will be trained on the correct locations for each TEA device and will receive an additional 4 weeks of treatment with the device.

Note: The gastric emptying breathalyzer test (GEBT) was removed, and the two-day visits were shortened to one-day to improve patient recruitment and retention.

ELIGIBILITY:
Inclusion Criteria:

* At least a 3-month history of diabetic gastroparesis symptoms on an on-going basis; at least one severe gastroparetic symptom or two moderate gastroparetic symptoms (e.g. vomiting, nausea, early satiety, bloating, or epigastric or abdominal pain) during the screening.
* Documented delayed gastric emptying within past 3 years
* Stable concomitant medications, defined as no changes in regimen for at least 2 weeks prior to the experiment (daily adjustments of insulin doses are permitted if patient has diabetes)

Exclusion Criteria:

* Currently receiving parenteral feeding or presence of a nasogastric or other enteral tube
* History of gastric surgery such as fundoplication, gastrectomy, or vagotomy
* Symptoms suggestive of gastroparesis with no diagnosis of diabetes
* Pregnancy or expect to conceive during the course of the study
* Uncontrolled diabetes mellitus (HbA1c > 11%).
* Having any implanted medical device, such as cardiac pacemaker or Entera device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Change in American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptoms Index-Daily Diary (ANMS GCSI-DD) | From baseline to up to 84 days
  A 24-hours recall period and five symptoms related to delayed emptying from the stomach: nausea, early satiety, postprandial fullness, upper abdominal pain, and vomiting.
  Scoring of ANMS GCSI-DD: The severity scores of four gastroparesis-related symptoms (nausea, early satiety, postprandial fullness, upper abdominal pain) range from 0-none to 4-very severe. Vomiting frequency is scored as 0 episodes, 1 episode, 2 episodes, 3 episodes or 4 or more episodes (capped as 4). The ANMS GCSI-DD total gastroparesis symptom daily score is generated by summing the scores on each of the five symptom items (nausea, early satiety, postprandial fullness, upper abdominal pain, and number of vomiting episodes) and then dividing by 5, that is the number of items within the gastroparesis related symptom score. Thus, the minimum score is 0 and the maximum score is 4. Higher numbers indicate greater symptom impact.
  Scores will be compared from day 0 to day 84.

SECONDARY OUTCOMES:
36-Item Short Form Survey Instrument (SF-36) to measure quality of life (QOL) | 8 weeks
  A 36 question assessment to score overall quality of life. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Gastric accommodation | 8 weeks
  A liquid nutrient drink test will be performed during which the patient will be asked to drink at a speed of 60ml/min until reaching the maximum tolerable volume (MTV). The postprandial symptoms of dyspepsia will be assessed at 10 , 20 and 30 min after completing the drink test with the patient scoring symptoms of bloating, fullness, nausea and pain using a visual analogue scale (VAS) with 100 mm lines and the words "unnoticeable" (0 mm) and "unbearable" (100mm) at each end. The sum of the four 100 mm visual analogue scales for each symptom provides an aggregate symptom score, the higher the score the greater the disability.
  A baseline test will be performed at visit 1.
Electrogastrogram (EGG) | Visit 1 and visit 2 at 8 weeks
  An EGG will be performed twice at both the baseline and at the 8 week visit. One 30-minute EGG will be performed prior to the gastric accommodation test and one 30-minute EGG will be performed after the nutrient drink test. The goal is to measure gastric slow waves. The difference in slow waves will be compared pre- and post- gastric accommodation. Slow waves will also be compared between visit 1 and visit 2
Electrocardiogram (ECG) | Visit 1 and visit 2 at 8 weeks
  An ECG will be performed twice at both the baseline and at the 8 week visit. One 30-minute ECG will be performed prior to the gastric accommodation test and one 30-minute EGG will be performed after the nutrient drink test. The goal is to measure autonomic function via calculating the heart rate variability (HRV). The difference in HRV will be compared pre- and post- gastric accommodation. HRV will also be compared between visit 1 and visit 2

OTHER OUTCOMES:
36-Item Short Form Survey Instrument (SF-36) to measure quality of life (QOL) | 12 weeks
  A 36 question assessment to score overall quality of life. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Borko Nojkov, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared. However, the study protocol and the study results will be shared

REFERENCES:
- [Background] Ma D, Han JS, Diao QH, Deng GF, Ping XJ, Jin WJ, Wu LZ, Cui CL, Li XD. Transcutaneous electrical acupoint stimulation for the treatment of withdrawal syndrome in heroin addicts. Pain Med. 2015 May;16(5):839-48. doi: 10.1111/pme.12738. PMID 25989154
- [Background] Jiang Y, Liu J, Liu J, Han J, Wang X, Cui C. Cerebral blood flow-based evidence for mechanisms of low- versus high-frequency transcutaneous electric acupoint stimulation analgesia: a perfusion fMRI study in humans. Neuroscience. 2014 May 30;268:180-93. doi: 10.1016/j.neuroscience.2014.03.019. Epub 2014 Mar 20. PMID 24657460
- [Background] Qu F, Wang FF, Wu Y, Zhou J, Robinson N, Hardiman PJ, Pan JX, He YJ, Zhu YH, Wang HZ, Ye XQ, He KL, Cui L, Zhao HL, Ye YH. Transcutaneous Electrical Acupoint Stimulation Improves the Outcomes of In Vitro Fertilization: A Prospective, Randomized and Controlled Study. Explore (NY). 2017 Sep-Oct;13(5):306-312. doi: 10.1016/j.explore.2017.06.004. Epub 2017 Jun 30. PMID 28915981
- [Background] Yu Y, Wei R, Liu Z, Xu J, Xu C, Chen JDZ. Ameliorating Effects of Transcutaneous Electrical Acustimulation Combined With Deep Breathing Training on Refractory Gastroesophageal Reflux Disease Mediated via the Autonomic Pathway. Neuromodulation. 2019 Aug;22(6):751-757. doi: 10.1111/ner.13021. Epub 2019 Jul 26. PMID 31347247
- [Background] Zhang B, Xu F, Hu P, Zhang M, Tong K, Ma G, Xu Y, Zhu L, Chen JDZ. Needleless Transcutaneous Electrical Acustimulation: A Pilot Study Evaluating Improvement in Post-Operative Recovery. Am J Gastroenterol. 2018 Jul;113(7):1026-1035. doi: 10.1038/s41395-018-0156-y. Epub 2018 Jun 21. PMID 29925916

DOCUMENTS (1):
  • Informed Consent Form (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT05362578/ICF_000.pdf